CLINICAL TRIAL: NCT00583102
Title: A Dose Escalation Phase I/II Study of Lovastatin With High-Dose Cytarabine for Patients With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Dose Escalation Phase I/II Study of Lovastatin With High-Dose Cytarabine for Refractory or Relapsed AML
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual, PI left institution
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Raymond J Hohl, Professor Emeritus, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200104050
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; Lovastatin; Cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lovastatin followed by Cytarabine (Experimental): The subject will receive high dose cytarabine as well as lovastatin. The subject will take doses of lovastatin twice a day, about 12 hours apart. On the third day, the subject will begin high-dose cytarabine IV over 3 hours, twice a day, starting 1 hour after the lovastatin dose for 5 days.
  Interventions: Drug: Cytarabine; Drug: Lovastatin

INTERVENTIONS:
Drug: Cytarabine — Cytarabine dosage: 3.0 g/m2 IV over 3 hours every 12 hours on days 3-7.
  Other Names: CYTOSAR-U; Depocyt
Drug: Lovastatin — Lovastatin dosage: The first dose level will be lovastatin at 0.5 mg/kg/day. After each patient reaches day 14 subsequent patients will be treated at incrementally increasing doses that are 1 mg/kg/day, 2 mg/kg/day, 4 mg/kg/day, 8 mg/kg/day, 12 mg/kg/day, 18 mg/kg/day, and 24 mg/kg/day. If MTD is not reached at this dose of 24 mg/kg/day further dose escalations will occur with a 33% increase in dose at each level rounded to the nearest mg/kg/day.
  Other Names: Mevacor; Altoprev

SUMMARY:
The purpose of this study is to test the safety and effectiveness of combining a drug known as Lovastatin to the chemotherapy drug cytarabine. Lovastatin is currently used to lower blood cholesterol levels and lab data suggests that it increases the anti-leukemia activity of cytarabine. This research is being done because high doses of cytarabine induce remissions in only about 25% of patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
The rationale for combining lovastatin with cytosine arabinoside (HiDAC) in this trial is based on a study in press in Leukemia Research. This study demonstrated that there are synergistic interactions between cytosine arabinoside and lovastatin against human leukemia cell lines. In particular, this synergistic activity was observed in MTT assay. Given that there is such synergistic interaction in vitro it is reasonable to determine whether such interaction occurs in vivo. The proposed trial thus uses standard doses of HiDAC with incrementally increasing dose of lovastatin. This particular trial will follow an accelerated titration for lovastatin. The first dose level will be lovastatin at 0.5 mg/kg/day, divided into two daily PO doses given Q 12 hours on Days 1 -7 for a total of 14 doses. Doses should be rounded to the nearest 20 mg. After each subject reaches day 14, subsequent subjects will be treated at incrementally increasing doses that are 1 mg/kg/day, 2 mg/kg/day, 4 mg/kg/day, 8 mg/kg/day, 12 mg/kg/day, 18 mg/kg/day, and 24 mg/kg/day, with all doses divided into two daily PO doses given Q 12 hours on Days 1 - 7 for a total of 14. If MTD is not reached at the 24 mg/kg/day dose level, further dose escalations will occur with a 33% increase in dose at each level, rounded to the nearest 20 mg/kg/day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary refractory AML (that is no prior remission). Patients who have greater than 10% AML blasts in the bone marrow or blood upon recovery from two cycles of standard cytarabine- and anthracycline-based induction chemotherapy are eligible. Patients who have received etoposide and/or 6-thioguanine during remission induction will be eligible.
* Patients with relapsed AML. Patients must have had a documented remission lasting > 30 days at some point during their prior therapy. Their current relapse must be untreated. Relapse is defined as the presence of greater than 10% AML blasts in the bone marrow or blood after having had a documented remission.
* Patients who have received a high-dose cytarabine containing regimen (>2 g/m2/dose) within 3 months prior to registration on this protocol are not eligible.
* No active CNS involvement. A lumbar puncture prior to treatment is not required and should not be performed in the absence of significant CNS symptoms or signs.
* Non-pregnant and non-nursing. Treatment under this protocol would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective means of birth control.

Exclusion Criteria:

Although NOT considered formal Exclusion Criteria, study physicians are strongly encouraged as part of this decision-making process to recognize that the following may increase the risks to a subject entering this protocol:

* Other serious illnesses which would limit survival to <2 years, or a psychiatric condition which would prevent compliance with treatment or informed consent.
* Performance Status > 2.
* Uncontrolled or severe cardiovascular disease, diabetes, pulmonary disease, or infection, which in the opinion of the treating physician, would make this protocol treatment unreasonably hazardous for the patient.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and considered by their physician to be at less than 30% risk of relapse within one year.
* Patients who have received any investigational agent within the prior 4 weeks.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-06 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Hohl, MD, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lovastatin Followed by Cytarabine
Started | 23
Completed | 20
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Lovastatin Followed by Cytarabine
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 64.3 [45.6 to 81.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate
Description: The primary study end point will be complete remission rate.
  Complete Remission (CR):
  Complete remission is defined as the presence of all of the following:
  Peripheral Blood Counts (sustained > 30 days)
  * Absolute neutrophil count ³1500/ml.
  * Platelet count ³100,000/ml.
  * No leukemic blasts in the peripheral blood.
  * Transfusion independent for red cells and platelets. Bone Marrow
  * Cellularity >20% with maturation of all cell lines.
  * No Auer rods.
  * <5% blast cells. No extramedullary leukemia (such as CNS or soft tissue involvement). OR Complete Response with Incomplete Platelet Recovery (CRp): CRp satisfies all CR criteria except platelets < 100,000/µL.
  Partial Remission (PR):
  Must meet all criteria of a CR except that the bone marrow may contain 5-24% blasts.
  Treatment Failure:
  Failure to achieve a CR.
Time Frame: 5 weeks
Population: 7 patients out of the 20 who completed the trial were primary refractory AML, so as per protocol these patients were not included for assessment and the early stopping rule.
Measure: Count of Participants; unit: Participants
Arm/Group | Lovastatin Followed by Cytarabine
Number analyzed (Participants) | 13
Participants
  Complete Remission(CR) | 7
  Partial Remission(PR) | 3
  Treatment Failure | 3

ADVERSE EVENTS:
Groups:
- Lovastatin Followed by Cytarabine: The subject will receive high dose cytarabine as well as lovastatin. The subject will take doses of lovastatin twice a day, about 12 hours apart. On the third day, the subject will begin high-dose cytarabine IV over 3 hours, twice a day, starting 1 hour after the lovastatin dose for 5 days.
  Lovastatin and Cytarabine: Cytarabine dosage: 3.0 g/m2 IV over 3 hours every 12 hours on days 3-7.
  Lovastatin dosage: The first dose level will be lovastatin at 0.5 mg/kg/day. After each patient reaches day 14 subsequent patients will be treated at incrementally increasing doses that are 1 mg/kg/day, 2 mg/kg/day, 4 mg/kg/day, 8 mg/kg/day, 12 mg/kg/day, 18 mg/kg/day, and 24 mg/kg/day. If MTD is not reached at this dose of 24 mg/kg/day further dose escalations will occur with a 33% increase in dose at each level rounded to the nearest mg/kg/day.
Arm/Group | Lovastatin Followed by Cytarabine
All-Cause Mortality (participants affected / at risk) | 6/23
Serious Adverse Events (participants affected / at risk) | 10/23
Other Adverse Events (participants affected / at risk) | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovastatin Followed by Cytarabine (N=23)
Cardiac left ventricular function (Cardiac disorders) | 1 (1)
Cardiac troponin T (cTnT) (Cardiac disorders) | 1 (1)
Fibrinogen (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 1 (1)
Hypokalemia,Hypophosphatemia,elevated ALT (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Elevated GGT (Hepatobiliary disorders) | 1 (3)
Decreased WBCs, Grade 3 lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Decreased albumin (Blood and lymphatic system disorders) | 1 (1)
Pneumonia infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Stroke (Cardiac disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Candidemia (Infections and infestations) | 1 (1)
Thrombosis/embolism (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovastatin Followed by Cytarabine (N=23)
Nausea (Gastrointestinal disorders) | 6 (10)
Emesis (Gastrointestinal disorders) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 5 (5)
Fatigue (General disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Thumb numbness (Nervous system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (3)
c-difficile infection (Gastrointestinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Edema (Cardiac disorders) | 3 (3)
GI bleed (Gastrointestinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fluid overload (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Bilirubin (Hepatobiliary disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7)
Enlarged gall bladder (Gastrointestinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Weight gain (General disorders) | 4 (4)
Elevated Alkaline Phosphate (Metabolism and nutrition disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Decreased white blood cell count (Blood and lymphatic system disorders) | 5 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Insomnia (General disorders) | 2 (2)
Hemorrhage (Picc site) (Injury, poisoning and procedural complications) | 1 (1)
Oral pain (General disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (6)
Elevated alanine transaminase (ALT) (Metabolism and nutrition disorders) | 4 (4)
Elevated aspartate transaminase (AST) (Metabolism and nutrition disorders) | 4 (4)
Elevated glucose (Metabolism and nutrition disorders) | 4 (4)
Klebsiella oxytoca (Infections and infestations) | 1 (1)
Decreased calcium (Metabolism and nutrition disorders) | 2 (2)
Decreased hemoglobin (Blood and lymphatic system disorders) | 4 (4)
Decreased platelets (Blood and lymphatic system disorders) | 4 (4)
Increased Prothrombin time (PTT) (Blood and lymphatic system disorders) | 2 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 1 (1)
Decreased lymphocytes (Blood and lymphatic system disorders) | 2 (2)
Decreased sodium (Metabolism and nutrition disorders) | 1 (1)
Decreased magnesium (Metabolism and nutrition disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Diaphoretic (General disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Oral lesion (General disorders) | 1 (1)
Jaw/tooth pain (General disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Decreased bicarbonate (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
White patch on tongue (General disorders) | 1 (1)
Oral infection, herpes simplex Type I (Infections and infestations) | 1 (1)
T-spine nodule (Musculoskeletal and connective tissue disorders) | 1 (1)
Deep Vein Thrombosis, upper extremity (Vascular disorders) | 1 (1)
Difficulty swallowing (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Toothache (Infections and infestations) | 2 (2)
Infection, c-diff (Infections and infestations) | 1 (1)
Pain, bone marrow biopsy site (Injury, poisoning and procedural complications) | 1 (1)
Neurological, poor finger-nose touch (Nervous system disorders) | 1 (1)
Pain, right thigh (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis, left hand (Skin and subcutaneous tissue disorders) | 1 (1)
Pain, right groin (Musculoskeletal and connective tissue disorders) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (2)
Pain, suprapubic (Renal and urinary disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Neutropenia (General disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
T-spine wound discomfort (Injury, poisoning and procedural complications) | 1 (1)
Weight loss (General disorders) | 3 (3)
Oral thrush (Infections and infestations) | 2 (2)
Increased GGT (Metabolism and nutrition disorders) | 2 (2)
Infection with neutropenia (e-coli) (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Neutropenic fever (Infections and infestations) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Decreased leukocytes (Blood and lymphatic system disorders) | 2 (4)
Decreased ANC (Blood and lymphatic system disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Increased troponin t (Cardiac disorders) | 1 (1)
Cardiac ventricular function (Cardiac disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1)
Headache (General disorders) | 1 (2)
Pain at new hickman line site (Injury, poisoning and procedural complications) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (2)
Neutrophils (Blood and lymphatic system disorders) | 1 (2)
Abscessed tooth, infection (Infections and infestations) | 1 (1)
Thrombocytropenia (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Increased creatinine (Metabolism and nutrition disorders) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial terminated early due to slow accrual. PI left the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes